CLINICAL TRIAL: NCT02987075
Title: A Comparison of Ongoing Pregnancy Rate Between Cleavage Stage and Early Compacting Embryo Transfer at 66±2 Hours After ICSI Using Single Step Culture Medium
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Vietnam National University (Other)
Responsible Party: Principal Investigator, Manh Tuong Ho, Director, Vietnam National University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCKH-08-2016
Record Dates: First submitted 2016-11-25; First posted 2016-12-08 (Estimated); Last update posted 2017-07-17 (Actual); Status verified 2017-07

CONDITIONS: Infertility
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Early compaction embryo group (Other): patients have compacting embryos at 66±2 hours after ICSI
  Interventions: Other: Compacting embryo transferring
- Cleavage stage embryo group (Other): patients have non-compacting embryos with 7-9 cells, under 20% fragmentation. at 66±2 hours after ICSI
  Interventions: Other: Non- compacting embryo transferring

INTERVENTIONS:
Other: Compacting embryo transferring — transfer of 2 utilizable compacting embryos
  Arms: Early compaction embryo group
Other: Non- compacting embryo transferring — transfer of 2 utilizable non-compacting embryos have 7-9 cells with under 20% fragmentation.
  Arms: Cleavage stage embryo group

SUMMARY:
A comparison of ongoing pregnancy rate between cleavage stage and early compacting embryo transfer at 66±2 hours after ICSI using single step culture medium

DETAILED DESCRIPTION:
A prospective cohort study to compare the outcomes of transferring the early compacting and the cleavage day 3 embryos.

All participants were treated with a gonadotropin-releasing antagonist protocol according to local protocol. Recombinant follicle stimulating hormone was given for five days starting on the second or third day of the menstrual cycle at a starting dose individualized for each participant as follows: 150, 225 or 300 IU/day, respectively, in participants with anti-Müllerian hormone levels of <2.1 ng/mL, 0.7-2.1 ng/mL or <0.7 ng/mL. This dosage could then be titrated based on clinical judgement of the investigator. Follicular development was monitored using ultrasound scanning and measurement of estradiol and progesterone levels, starting on day five of stimulation; scanning and hormonal measurements were repeated every two to three days, depending on follicle size. An antagonist was routinely used on day five until the day of human chorionic gonadotropin administration. Criteria for administration of recombinant human chorionic gonadotropin (5,000 IU) was the presence of at least two leading follicles of 17 mm in diameter. Oocyte retrieval was performed 36 hours after recombinant human chorionic gonadotropin administration.

Insemination was performed using intra-cytoplasmic sperm injection at three to four hours after oocyte retrieval; only matured oocytes were inseminated. Fertilization check was performed under inverted microscope at 16-18 hours after insemination. Embryo evaluation was performed on day 3 at fixed time point after fertilization (66±2 hours) using the Istanbul consensus. As a rule, two useful embryos are transferred in patients if having either early compaction or still on cleavage stage.

Early compaction embryo transfer group: transfer of 2 utilizable compacting embryos.

Cleavage stage embryo transfer group: transfer of 2 utilizable non-compacting embryos have 7-9 cells with under 20% fragmentation.

Embryo transfer was performed using a soft catheter by a standard technique under ultrasound guidance. Intensive luteal phase support was provided using progesterone gel and estradiol. At least 18 days after OPU, a urinary pregnancy test is performed. If the pregnancy test is positive, vaginal and/or abdominal ultrasonographic investigation is performed between 35 and 42 days (5 to 6 weeks) after ET to confirm a clinical pregnancy and at least 70 days (≥10 weeks) after ET to confirm an ongoing pregnancy.

Other clinical parameters will also be evaluated: serum hormone levels, fertilization rate, number and quality of day 3 embryos, implantation rate, ectopic pregnancy rate and miscarriage rate.

ELIGIBILITY:
Inclusion Criteria:

* IVF treatment for infertility
* Controlled ovarian hyperstimulation by GnRH antagonist protocol.
* IVF cycles ≤2
* Eligible for transfer of 2 embryos on day 3
* Have at least 2 embryos which are 7-9 cells and fragmentation ≤20%, that had either early compaction or still on cleavage stage

Exclusion Criteria:

* Oocyte donation cycles
* Abnormal uterine
* Using GnRH agonist for triggering.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 430 (Estimated)
Dates: Start 2016-12; Primary Completion 2017-11 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
The primary outcome measure was ongoing pregnancy rate, defined as a pregnancy with a detectable heart rate at 12 weeks of gestation or beyond. | 12 weeks

SECONDARY OUTCOMES:
Clinical pregnancy rate, defined as the presence of a gestational sac under ultrasonography | 7 weeks
Implantation rate (number of gestational sacs on ultrasound at 7 weeks / total number of embryos transferred x 100). | 7 weeks
Ectopic pregnancy rate, defined as the ectopic nidation of a pregnancy, confirmed with sonography or laparoscopy | 7 weeks
Miscarriage rate, defined as the loss of a pregnancy prior to 12 weeks gestation | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Tuong M Ho, MD, Principal Investigator — CGRH - Vietnam National University
Locations (1):
- My Duc Hospital, Ho Chi Minh City, Vietnam

IPD SHARING:
Plan to Share IPD: No